CLINICAL TRIAL: NCT01864590
Title: Open Abdomen: Vacuum Pack Versus Sylo Bag and Mesh Protocol - A Randomized Trial
Brief Title: Open Abdomen: Vacuum Pack Versus Sylo Bag and Mesh Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Carlos Hernando Morales, Chief Surgery Department, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University Of Antioquia
Record Dates: First submitted 2013-05-19; First posted 2013-05-29 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Open Abdomen; Temporary Abdominal Closure Mechanisms
Keywords: Open Abdomen; Negative Pressure Wound Therapy; Temporary Abdominal Closure; Mesh; Abdominal reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Abdomen - Vacuum Pack (Experimental): Patients that Require open abdomen
  Interventions: Device: Vacuum Pack
- Double Sylo Bag - Mesh Protocol (Active Comparator): Open Abdomen
  Interventions: Device: Double Sylo Bag - Mesh Protocol

INTERVENTIONS:
Device: Vacuum Pack — Vacuum Pack Technique described by Barker et al.
  Arms: Open Abdomen - Vacuum Pack
Device: Double Sylo Bag - Mesh Protocol — double sylo bag, one underneath the fascia and the other sutured to the skin, at the initial operation.
  At subsequent surgeries once the abdomen is clean the investigators leave the same subfascial sylo bag and use a prolene mesh attached to the fascia. This mesh is resutured every day until the abdominal fascia is approximated enough to permit closure
  Arms: Double Sylo Bag - Mesh Protocol

SUMMARY:
The open abdomen is a valid and accepted surgical tactic for the trauma and acute care patient. There have been many mechanisms described for its management, but the most accepted strategy is the vacuum pack. At our hospital the investigators have used for many years a double sylo bag, one underneath the fascia and the other sutured to the skin, at the initial operation. At subsequent surgeries once the abdomen is clean the investigators leave the same subfascial sylo bag and use a prolene mesh attached to the fascia. Every day the investigators try to tighten the mesh with sutures until the abdomen can be closed. This study´s objective is to compare our double sylo bag- mesh protocol with the vacuum pack to determine which is related to a higher fascial closure rate.

DETAILED DESCRIPTION:
The Investigators plan to compare our double sylo-mesh protocol with the vacuum pack technique described by Barker et al. To accomplish this they have designed a randomized trial that will include patients that require an open abdomen strategy according to their attending physician either due to a traumatic or a medical cause. Once the surgeon decides to leave the abdomen open, one of the nurses will pick up an envelope from the randomization box and read out loud the patients allocation (Vacuum pack or Double sylo bag-mesh protocol) . During subsequent surgeries the patient must continue with the same strategy for a minimum of 21 days or until fascial closure. The patients will be followed during their whole hospital stay to determine complication rates and fascial closures.

ELIGIBILITY:
Inclusion Criteria:

* Open Abdomen

Exclusion Criteria:

* Patients that die in the first 48 hours after the initial intervention

Ages: 13 Years to 96 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Fascial Closure Rate | Until hospital discharge Aprox 60 days

SECONDARY OUTCOMES:
Gastrointestinal Fistulas | Until hospital discharge Aprox. 60 days
Abdominal Abscess | Until hospital discharge Aprox. 60 days
Fascial Closure Dehiscence | Until hospital discharge Aprox. 60 days
Length of Stay | Until hospital discharge Aprox. 60 days
Day of Fascial Closure | Until hospital discharge Aprox. 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos H Morales, MD, Principal Investigator — Universidad de Antioquia
Locations (1):
- Hospital Universitario San Vicente Fundacion, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Correa JC, Mejia DA, Duque N, J MM, Uribe CM. Managing the open abdomen: negative pressure closure versus mesh-mediated fascial traction closure: a randomized trial. Hernia. 2016 Apr;20(2):221-9. doi: 10.1007/s10029-016-1459-9. Epub 2016 Feb 1. PMID 26833235